CLINICAL TRIAL: NCT00002096
Title: A Phase I Pharmacokinetic Study in HIV-Positive Subjects of Oral Ganciclovir and Concomitant Antiretroviral Zidovudine and Didanosine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 059E; ICM 1776
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1993-11

CONDITIONS: Cytomegalovirus Infections; HIV Infections
Keywords: Didanosine; Ganciclovir; Drug Interactions; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome; Zidovudine
MeSH Terms: conditions — Cytomegalovirus Infections; HIV Infections; Multiple Acyl Coenzyme A Dehydrogenase Deficiency; Acquired Immunodeficiency Syndrome | interventions — Zidovudine; Didanosine; Ganciclovir

INTERVENTIONS:
Drug: Zidovudine
Drug: Didanosine
Drug: Ganciclovir

SUMMARY:
To determine whether there is a pharmacokinetic drug interaction between oral ganciclovir and oral zidovudine (AZT) and between oral ganciclovir and oral didanosine (ddI). To determine whether concurrent administration of probenecid affects the pharmacokinetics of oral ganciclovir. To obtain data on the short-term safety of oral ganciclovir administered concurrently with AZT, ddI, or probenecid in HIV-positive patients.

DETAILED DESCRIPTION:
Patients currently on either AZT or ddI receive ganciclovir therapy.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Required:

* Concomitant AZT or ddI.

Allowed:

* Probenecid.
* Aerosolized pentamidine.

Patients must have:

* Asymptomatic HIV infection.
* CMV seropositivity or CMV culture positivity at present or at any time in the past.
* No history of CMV disease (e.g., retinitis, colitis) or any other AIDS-defining illness.
* Treatment with AZT or ddI for at least 1 month prior to study entry.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms and conditions are excluded:

* Uncontrolled diarrhea (three or more loose stools/day).
* Clinically significant gastrointestinal symptoms including persistent nausea or abdominal pain.
* AZT patients only:
* Deficiency in glucose-6-phosphate dehydrogenase.
* ddI patients only:
* Grade 2 or worse peripheral neuropathy.

Concurrent Medication:

Excluded:

* Combination antiretroviral therapy.
* G-CSF or GM-CSF.
* Acyclovir.
* Amphotericin B.
* Amikacin.
* Captopril.
* Carbamazepine.
* Cimetidine.
* Cyclosporine.
* Glutethimide.
* Gentamicin.
* Griseofulvin.
* Ibuprofen.
* Imipenem-Cilastatin.
* Lithium.
* Methicillin.
* Methotrexate.
* Naproxen.
* Pentamidine (Pentam 300) (Aerosolized drug permitted).
* Phenacetin.
* Phenobarbital.
* Phenytoin.
* Piroxicam.
* Ribavirin.
* Rifampin.
* Tobramycin.
* Vidarabine.
* Zalcitabine.
* Other investigational drugs.

Patients with the following prior conditions are excluded:

* History of hypersensitivity to acyclovir or ganciclovir.
* AZT patients only:
* History of gout, uric acid, kidney stones, peptic ulcer or porphyria.
* ddI patients only:
* History of pancreatitis or alcoholism, or seizures within 6 months prior to study entry or prior need for anticonvulsant therapy.

Prior Medication:

Excluded:

* Combination antiretroviral therapy within 1 month prior to study entry.

Required:

* AZT at 500 mg/day for at least 1 month prior to study entry (with 100 mg administered five times per day for at least 1 week prior to study entry). OR
* ddI at recommended dose for at least 1 month prior to study entry (with 250 mg administered every 12 hours for at least 1 week prior to study entry).

History of alcoholism (in ddI patients).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Ctr for Special Immunology, Irvine, California
  - Georgetown Univ Med Ctr, Washington D.C., District of Columbia
  - Univ TX Galveston Med Branch, Galveston, Texas

REFERENCES:
- [Background] Gaines K, Wong R, Jung D, Cimoch P, Lavelle J, Pollard R. Pharmacokinetic interactions with oral ganciclovir: zidovudine, didanosine, probenecid. Int Conf AIDS. 1994 Aug 7-12;10(1):7 (abstract no 004B)